CLINICAL TRIAL: NCT06576869
Title: "Timing Of Tourniquet Release, A Prospective Randomized Trial"
Brief Title: Timing of Tourniquet Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Brett Lewellyn, Principal Investigator, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22.028.02
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Injury
Keywords: Tourniquet study
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Closure without releasing the tourniquet. (Active Comparator): Tourniquet is dropped after closure.
  Interventions: Procedure: Upper extremity orthopedic surgeries.
- B: Releasing the tourniquet and then closing the incision (Active Comparator): Tourniquet is dropped prior to closure.
  Interventions: Procedure: Upper extremity orthopedic surgeries.

INTERVENTIONS:
Procedure: Upper extremity orthopedic surgeries. — Upper extremity orthopedic surgeries that require the use of a tourniquet.

SUMMARY:
This will be a prospective randomized clinical trial comparing clinical outcome measures in patients who undergo elective upper extremity surgery when tourniquet is dropped prior to closure as opposed to when tourniquet is dropped after closure. The study will compare objective data obtained intraoperatively as well as standard clinical outcome measures such as pain scores at routine follow up.

DETAILED DESCRIPTION:
Patients will be enrolled prior to surgery and consented to participate in the study [HPJ2]. Patients will be enrolled by the research staff with a provider including attending and resident surgeons as well as advanced practiced providers that are assigned to the upper extremity team. A computerized random number generator will be used to randomize patient allocation to either study arm: closure without releasing the tourniquet vs releasing the tourniquet and then closing the incision. Randomization will occur at the time of surgery. In order to standardize the procedure a 4-inch ace wrap will be wrapped around the upper arm and a tourniquet will be placed over this in order to ensure adequate padding [HPJ3] [AW4]. At the conclusion of the surgical procedure but prior to skin closure, the randomized number will be revealed to the surgeon and the surgeon will either release the tourniquet or will keep the tourniquet inflated and then close the skin. After the surgery is completed, information will be collected on the intraoperative data collection form to include: • Length and exact location of incision• Whether the patient is on anticoagulant medication., o This includes type/dose of medicationo Duration for taking the medicationo Was the medication halted prior to surgery; if so, when• Surgeon performing the surgery• Surgical procedure• Surgery location (Ambulatory Care Center (ACC), Orlando Regional Medical Center (ORMC), etc.) • When tourniquet is dropped (before/after closure)• Tourniquet Time• Time from tourniquet release to closure• Total Surgical time (time from incision until complete skin closure) • Turnover time• Was electrocautery required to control any bleeding; if so, what type and what was electrocauterized? Clinical outcome measures collected during postoperative follow up. • Visual analog pain scale• Quick Disability of the Arm, Shoulder and Hand (DASH) form• Complications including hematoma size• Satisfaction with treatment (scale 1-5)o completely satisfied - 5, somewhat satisfied - 4, neither satisfied or dissatisfied - 3, partly dissatisfied - 2, completely dissatisfied - 1• Likely to recommend this surgery to a friend family member who has the same condition - yes or no Patients enrolled in the study will follow up in clinic at the following time intervals: 2 weeks, 10 weeks, and 6 months per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Consented study subjects 18 years or older
* Subjects with any upper extremity injury or ailment that would require the use of a tourniquet while doing surgery
* Subject undergoing surgery by one of the six fellowship trained Orlando Health upper extremity surgeons previous listed
* Subject without prior surgery to the operative extremity

Exclusion Criteria:

* Subject under the age of 18 at the time of consent/enrollment
* Subject has had previous surgical procedures at the surgery site
* Subject with bleeding disorder comorbidities
* Subjects who have tourniquet released and then re-inflated during their procedure
* Subjects who do not have English as their preferred language and require an interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Visual analog pain scale | 2 weeks, 10 weeks and 6 months.
  Visual number scale to rate pain from 0-10 where 0 equals no pain and 10 equals worst possible pain
Quick DASH form | 2 weeks, 10 weeks, 6 months.
  Assessment of symptoms and ability to perform certain activities.
Hematoma assessment | 2 weeks, 10 weeks, 6 months.
  Performed by MD, assessment of the presence of a hematoma and if present, it is measured.
Satisfaction with surgery | 2 weeks, 10 weeks, 6 months.
  Patient to rate their satisfaction with their surgery and to indicate whether or not they would recommend the surgery to family/friends with the same condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health Jewett Orthopedic Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
In order to protect the rights of our study participants, protected heath information will not be identified or shared.

REFERENCES:
- [Background] Zhang P, Liang Y, He J, Fang Y, Chen P, Wang J. Timing of tourniquet release in total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Apr;96(17):e6786. doi: 10.1097/MD.0000000000006786. PMID 28445317
- [Background] Fitzgibbons PG, Digiovanni C, Hares S, Akelman E. Safe tourniquet use: a review of the evidence. J Am Acad Orthop Surg. 2012 May;20(5):310-9. doi: 10.5435/JAAOS-20-05-310. PMID 22553103
- [Background] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159